CLINICAL TRIAL: NCT00294749
Title: Comparison Between Short and Long Schemes of Antibiotic Prophylaxis for Transrectal Prostate Biopsy. A Multicentre Prospective Randomised Study
Brief Title: Short or Long Schemes of Antibiotic Prophylaxis for Prostate Biopsy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2005-005959-17
Record Dates: First submitted 2006-02-19; First posted 2006-02-22 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Men Who Must Undergo a Prostate Biopsy Related to Prostate Cancer Suspicion.
Keywords: Prostate,; Infection,; Biopsy,; Antibiotic,; Prophylaxis
MeSH Terms: conditions — Infections | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ciprofloxacine

SUMMARY:
The purpose of this study is to determine whether long antibiotic prophylactic is more effective than a short traitement in infective complications for prostate biopsy

DETAILED DESCRIPTION:
Prophylactic antibiotic is used to minimize the infective complications risk following transrectal biopsy of the prostate.

The majority of works points to the need of antibiotic prophylaxis previously to transrectal prostate biopsy. However, there is a lot of controversy and diversity of therapeutic schemes in the literature concerning the ideal drug to be used and the time employed for infectious prophylaxis.

The objective of this randomised study was to assess 2 different schemes of antimicrobial prophylaxis, aiming to determine the difference in infective complications with a single dose of ciprofloxacin 2 hours before the procedure vs. ciprofloxacin for 3 days

ELIGIBILITY:
Inclusion Criteria:

* abnormal digital rectal examination
* abnormal PSA values

To be excluded those patients with:

* ciprofloxacine contraindication
* indwelling urethral catheter,
* positive urine culture,
* presence of cardiac valve prosthesis,
* uncontrolled diabetes mellitus,
* use of antimicrobials in the 7 days prior to biopsy.
* Urinary endoscopic procedure in the 7 days prior to biopsy
* coagulation defect
* Renal insufficiency
* Hepatic insufficiency

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-02; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Bacteriuria five days after prostate biopsy

SECONDARY OUTCOMES:
- Clinically diagnosed infectious complications
- Other complications related to the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Irani Jacques, professor, Principal Investigator
Locations (1):
- Poitiers Hospital University, Poitiers, France